CLINICAL TRIAL: NCT00364312
Title: Improving Control With Activity and Nutrition
Brief Title: Lifestyle Interventions for Long Term Diabetes Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R18DK062942 (NIH)
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Type 2 Diabetes
Keywords: behavior therapy; dietary control; exercise; diabetes mellitus; behavior modification; blood glucose; clinical trial; diabetes education; health behavior; health care service utilization; obesity; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus; Health Behavior; Patient Acceptance of Health Care; Obesity | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: diet and physical activity

SUMMARY:
Lifestyle interventions have been shown to reduce heart disease risk and improve blood sugar control in clinical trials. This project will investigate whether those lifestyle interventions can be implemented long-term, in usual practice settings, by using dietitian case managers to coordinate lifestyle change in cooperation with fitness instructors and primary care clinicians.

DETAILED DESCRIPTION:
The proposed randomized trial investigates the effectiveness of lifestyle case management to encourage long-term lifestyle modifications in diet and physical activity, improve control of type 2 diabetes, reduce risk factors for progression of type 2 diabetes and cardiovascular disease, and improve quality of life, among health plan enrollees with type 2 diabetes and obesity. Patients agreeing to participate are randomly assigned to one of two conditions: 1) lifestyle case management, in which initial 12 month intensive diet and physical activity intervention is followed by 30 months of active maintenance directed by dietitians and physical trainers (the "lifestyle case management" group); 2) lifestyle intervention, in which there is no formal maintenance following the intensive lifestyle intervention (the "lifestyle intervention" group). Because the lifestyle case management intervention incorporates the content of the lifestyle intervention, we will be able to assess the incremental effectiveness of providing post-intervention lifestyle case management on glycemic control, cardiovascular risk, body composition, diet and physical activity habits, and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* treated for type 2 diabetes within one year prior to their entry into the trial, have a BMI at or above 30, and are 18 years of age or older

Exclusion Criteria:

* 1) end-stage renal disease (defined as being on dialysis), 2) active foot ulcers or infections (defined as an open wound or requiring drug therapy), 3) pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer) that precludes diet and physical activity changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2004-05; Study Completion 2009-12

PRIMARY OUTCOMES:
HbA1c
Waist circumference
Body mass index
Lipids
Health care utilization
Quality of life

SECONDARY OUTCOMES:
Diet
Physical activity
Diabetes knowledge
Social support
Self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Viktor E Bovbjerg, PhD MPH, Principal Investigator — University of Virginia; Jayne Q Crowther, RN MSN, Study Director — University of Virginia
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States